CLINICAL TRIAL: NCT04767399
Title: Comparison of Postoperative Pain After Root Canal Preparation, in Single and Multiple Visits, With Reciprocating and Rotary Single-File Systems: A Randomized Clinical Trial.
Brief Title: Comparison of Postoperative Pain After Instrumentation in Different Visits With Different Single File Systems.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Yahia Abdullah Alyami, postgraduate resident, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FPGRP/2020/497
Record Dates: First submitted 2021-02-12; First posted 2021-02-23 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single visit (Experimental): root canal treatment will be done in one visit
  Interventions: Behavioral: protaper next
- multiple visit (Experimental): root canal treatment will be done in multiple visit
  Interventions: Behavioral: protaper next

INTERVENTIONS:
Behavioral: protaper next — rotary systems used on patients need root canal treatment
  Other Names: Edge-one fire

SUMMARY:
Comparison of Postoperative Pain after Root Canal preparation, in Single and Multiple Visits, with Reciprocating and Rotary Single-File Systems: A Randomized Clinical Trial.

Aim:1. Compare between the postoperative pain after root canal preparation, in single and multiple visits.

2. To assess the influence of reciprocating and rotary single-file systems instrumentation on post-operative pain.

DETAILED DESCRIPTION:
Subjects allocation and randomization method:

* All diagnoses and treatment procedures will be performed by a single operator in one visit or multiple visits to eliminate or minimize individual variability in the treatment between clinicians.
* Total of 160 patients, as per the inclusion criteria will be intervened. This will be divided into two groups as follows:

  1. Group A (n=80) single visit.
  2. Group B (n=80) multiple visits.
* Group A and B will be subdivided into two groups (each group=40) based on the motion of the files to be used either Reciprocation EOF (Edge one Fire file) or Rotational motion PN (ProTaper Next files). Each subgroup will be divided based on either the tooth is vital or non-vital (each subgroup=20) as shown in study design (Figure 1).

(Figure 1)

* A pulpal and periapical diagnoses will be done for each tooth on taking careful history, clinical and radiographic examination based on the American Association of Endodontists (AAE 2008) diagnostic guidelines.
* The treatments in groups A or B by ProTaper Next or Edge one Fire will be randomized with sequentially numbered opaque sealed envelopes (SNOSE) with 40 patients in PN group and 40 patients in EOF group with allocation sequence and assigning to intervention which will be done by blinded second investigator at the time of cleaning and shaping, concealed from operator to reduce bias.

2.3. Treatment protocol Endodontic therapy consisted of local anesthesia (2% lidocaine with epinephrine 1:100,000 (Xylocaine; Dentsply Pharmaceutical, York, PA) administration and rubber dam isolation followed by access cavity preparation. A size # 10 stainless steel hand K-file (Dentsply) will be used to check the patency of canal. Root ZX II apex locator (J Morita Corp, Kyoto, Japan) will be used to determine the working length which will further confirmed using periapical radiographs After working length determination, the canal will be enlarged to size # 15 using stainless steel hand K-files (Dentsply). At this stage, randomization will be carried out by second investigator based on SNOSE method and patients will be assigned to two different rotary systems, namely, PN and EOF for cleaning and shaping. The patient will be blinded to the type of rotary system used for cleaning and shaping.

Systems Used for Cleaning and Shaping:

Reciprocating motion single file system (n=40): The canals in this group will be instrumented with an engine driven reciprocation motion using an Edge one Fire files (EOF) (EdgeEndo, Albuquerque, New Mexico) with the same preset program specific for the WaveOne Gold instruments, because Edge One Fire has no preset motion and manufacturer declare its full compatibility with WOG counter-clock wise reciprocating motion with an engaging angle of 150° and a disengaging angle of 30° at 300 rpm using an X-Smart Plus endodontic motor (Dentsply Maillefer) with S (20 .06) or P (25 .06) for narrow or severely curved canals and M (35 .04) or L (45 .03) for wide canals.

Rotation motion multiple file system (n=40): The canals in this group will be instrumented with an engine driven rotational motion using a ProTaper Next (PN, Dentsply Sirona Endodontics, Ballaigues, Switzerland) in continuous rotary motion at the speed of 300 rpm and torque 2 Ncm with X1 (17 0.4) and X2 (25 0.6) used for preparation of narrow and curved canals, using X3 (30 0.6), X4 (40 .06) and X5 (50 .06) for wide canals.

Irrigation Protocol:

The same irrigation protocol will be applied in all groups; 2.5% sodium hypochlorite (NaOCl) will be delivered using disposable syringes and a 31-G side-vented needle (NaviTip needle; Ultradent Products Inc, South Jordan, UT) inserted into the canal 3 mm short of the WL between each instrument change. A total of 25 mL 2.5% NaOCl will be delivered per canal. The smear layer formed during chemo-mechanical preparation will be removed by rinsing the canal with 1 mL 17% EDTA and leaving the canal filled with this solution for 1 minute. Patency of the apical foramen will be maintained during all the techniques by introducing a #10 or #15 K-type file (Dentsply) to a point 1 mm beyond the WL at each instrument change. The root canals will be thoroughly dried with paper points after irrigation and before obturation.

Obturation Techniques:

The canals will be subsequently filled with the gutta-percha cones of the respective systems and AH-plus sealer (Dentsply Maillefer) using the continuous wave of condensation technique ??? Excess gutta-percha will be removed with hot instrument and the coronal gutta-percha was vertically condensed. The gutta-percha level will be reduced using hot plugger to a depth of 2 mm from the CEJ.

The access cavity will be closed by Cavit and GIC

2.4. Assessment of post-operative pain and statistical analysis All the participants will be received a card containing VAS (visual analogue scale) to assess pain levels after root canal treatment at 12 h, 24 h and 48 h. According to this scale, the level of pain will be documented in the range of 0-10 numerically and verbally as no pain (0), mild pain (1, 2), moderate pain (3-5), sever pain (6, 7), very severe pain (8), and worst pain possible (9, 10). All the participants will be explained about the scale verbally before the start of the procedure.

Patients will be contacted over telephone by the same clinician at 12, 24 and 48 h time periods and ask to describe the general feeling in the area of the treated tooth, the presence, absence, and intensity of the pain numerical and verbal, and intake of analgesics if any. The information so obtained will be recorded at each follow-up period. None of the patients will be prescribed with medication immediately after the treatment. They will be asked to call the clinician by telephone if they feel any discomfort in the treated area at any point of the follow-up time. If patient complained of pain, then the clinician will prescribe ibuprofen 400 mg as over-the-counter drug.

Data Analysis: Responses of participants to the visual analogue scale and verbal pain scale will be entered into a data spreadsheet software. Differences in post-operative pain between different instruments and different visits will be analyzed using a combination of parametric and non-parametric inferential analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* a. All permanent teeth diagnosed with vital or non-vital pulps and need nonsurgical root canal treatment.

  b. Symptomatic, Asymptomatic maxillary and mandibular teeth with apical radiolucency c. All males and females with age between 19 to 60 years.

Exclusion Criteria:

* a. Teeth with Previously treated b. Teeth need surgical treatment. c. Primary teeth. d. Patients with sinus tract, periapical abscess and who had previously medications.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-09-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 24 months
  appointment treatment at 24 month [ Time Frame: 12, 24, 48, h ] where 0 out of 10 scale will indicates no pain and 10 out of 10 indicates worse pain

SECONDARY OUTCOMES:
Verbal analogue scale | 24 moths
  appointment treatment at 24 month [ Time Frame: 12, 24, 48, h ] where 0 out of 10 scale will indicates no pain and 10 out of 10 indicates worse pain

CONTACTS AND LOCATIONS:
Locations (1):
- Yahia Abdullah Alyami, Riyadh, Saudi Arabia